CLINICAL TRIAL: NCT01300559
Title: Efficacy of the TissueLink Coagulation System in Reducing Hemoglobin Loss During Multi-Level Spine Surgery
Brief Title: TissueLink Study During Multi-Level Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Salient Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00016175
Record Dates: First submitted 2011-02-03; First posted 2011-02-21 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-01

CONDITIONS: Low Back Pain
Keywords: efficacy; hemoglobin; spine
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Tissuelink device plus Unipolar electrocautery will be used in this arm of the study.
  Interventions: Device: Tissuelink device
- No treatment (No Intervention): Unipolar electrocautery without Tissuelink device will be used in this arm of the study.

INTERVENTIONS:
Device: Tissuelink device — Tissuelink device plus Unipolar electrocautery
  Other Names: Aquamantys
  Arms: Treatment Group

SUMMARY:
The overall objective of the investigators research is to test the clinical efficacy of the TissueLink™ (Salient Surgical Technologies, Inc.) coagulation system in minimizing hemoglobin loss intraoperatively. This is a prospective, randomized investigation that will be performed at Duke University Medical Center (DUMC). The overall goal of this study is to evaluate the efficacy of Tissue Link HemoSealing system in minimizing hemoglobin loss preoperatively, intraoperatively and postoperatively for patients undergoing multilevel elective spinal surgery. Not greater than eighty patients scheduled for elective, multi-level decompression and fusion spinal surgery with Dr. William Richardson will be randomized into two groups. Unipolar electrocautery will be used for intraoperative coagulation in one group and the Tissuelink device plus Unipolar electrocautery in the other. These are frequently performed cases with significant blood loss but otherwise low morbidity/mortality that would benefit from more effective intraoperative coagulation.

DETAILED DESCRIPTION:
Very little research exists in the use of TissueLink HemoSealing device in spinal surgery. One retrospective study by Snyder et al evaluated hemostatic efficacy of this technology in children undergoing surgery for spinal fusion and instrumentation. Although the study reported no statistically significant difference in transfusion rates, there was a reduction in amount of blood transfused and operative time which was attributed to hemostatic efficacy in comparison with conventional wound management during surgery. The surgeons also reported a clearer operative field, improving visualization during surgery. Finally, the reduction in operative time which they suggested might be due to the use of this new device may reduce other complications by diminishing overall anesthesia exposure and blood product transfusions. From this initial retrospective study, the authors concluded that the use of the TissueLink HemoSealing device in spine surgery may be an effective tool in control of intra- and post-operative blood loss and may significantly reduce blood related and operative complications. More rigorous research needs to be done to evaluate the efficacy of the TissueLink HemoSealing device in hemostasis in the area of spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Sex: Both males and females will be included
* Patient has a Body Mass Index (BMI) <40
* Patient is willing and able to cooperate
* Patient is in stable health and cleared for surgery
* Patient is a candidate for elective multilevel posterior lumbar compression and fusion spinal surgery at least two or greater lumbar level involvement
* Patient has completed the Informed Consent Form

Exclusion Criteria:

* Patient is unable or unwilling to comply with the entire study protocol
* Patient has a previously diagnosed coagulopathy
* Patient has preoperative hemoglobin <11 g/dL
* Patient has a Prothrombin Time and International Normalized Ratio (PT/INR) >1.3
* Patient has a Partial Thromboplastin Time (PTT) >40
* Patient has a platelet count <100k
* Patients will also be excluded if taking non-aspirin medications producing a bleeding diathesis undetectable by screening labs such as clopidogrel or ticlopidine within seven days of surgery or valproic acid (associated with thrombocytopenia)
* Trauma patients are excluded
* Patient is a poor compliance risk, i.e., history of ethanol, drug abuse
* Severe cardiac disorder requiring special fluid management protocols
* Patients with acute myocardial infarction and/or acute angina
* Patient is on Plavix or other long term anti-coagulation including aspirin (ASA) or other nonsteroidal antiinflammatory drugs (NSAIDs) may be included provided their medications are discontinued a minimum of 7 days prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Hill, MD, Principal Investigator — Duke University; William J Richardson, MD, Study Chair — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Hill SE, Broomer B, Stover J, White W, Richardson W. Bipolar tissue sealant device decreases hemoglobin loss in multilevel spine surgery. Transfusion. 2012 Dec;52(12):2594-9. doi: 10.1111/j.1537-2995.2012.03649.x. Epub 2012 Apr 15. PMID 22500572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 adult patients (age ≥ 18 years) undergoing elective, multilevel, posterior lumbar decompression and fusion with Dr William Richardson were randomly assigned into two groups.
Pre-assignment Details: Enrollment started 10/09/2006 and enrollment completed 09/13/2010 with a total of 60 eligible subjects.
Period: Overall Study
Arm/Group | Treatment Group | No Treatment
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | No Treatment | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 13 | 12 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 62.6 (11.3) | 61.8 (10) | 62.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Measurement g/dl
Description: The primary hypothesis was that use of the Aquamantys coagulation system in addition to unipolar cautery results in less intraoperative Hb loss compared with unipolar cautery alone during multilevel spinal decompression and fusion surgery.Intraoperatively, shed blood will be collected into a Cell-saver device. Surgical sponges will be recovered in a container of citrated normal saline. Prior to processing the salvaged blood from the cell-saver device, hemoglobin concentration (g/dL) and volume (dL) of the salvaged blood will be measured, allowing calculation of hemoglobin loss in grams.
Time Frame: At the end of surgery
Population: Based on pilot data, it was estimated that 29 patients per group would provide 90% power with = 0.01 to distinguish such a difference between groups. Therefore, the randomized study was planned for 60 patients.
Measure: Mean (95% Confidence Interval); unit: hemoglobin g/dl
Groups:
- Treatment Group: Tissuelink device plus Unipolar electrocautery will be used in this arm of the study. Hemoglobin loss for the participants in this group will be measured in g/dl.
- No Treatment Group: Unipolar electrocautery without Tissuelink device will be used in this arm of the study. Hemoglobin loss for the participants in this group will be measured in g/dl.
Arm/Group | Treatment Group | No Treatment Group
Number analyzed (Participants) | 30 | 30
hemoglobin g/dl | 66.2 [14.4 to 174.1] | 102.4 [55.5 to 197.3]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Clinical assessment of subjects
Arm/Group | Treatment Group | No Treatment
Serious Adverse Events (participants affected / at risk) | 3/30 | 3/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=30) | No Treatment (N=30)
Serous wound drainage without evidence of infection. (Vascular disorders) | 1 (1) | 0 (0)
Dural tear. (Spinal tissue tear) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound hematoma. (bruise) (Vascular disorders) | 1 (1) | 0 (0)
Urinary tract infection. (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation. (Irregular heart beat) (Cardiac disorders) | 0 (0) | 1 (1)
Fever with a gout flare. (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
None encountered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less